CLINICAL TRIAL: NCT03236896
Title: Studying the Impact of Exercise on Hot Flashes Using Mobile Fitbit Flex, MENQOL Scale and Hot Flash Diary
Brief Title: Studying the Impact of Exercise on Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Sireesha Reddy, Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E14055
Record Dates: First submitted 2017-04-18; First posted 2017-08-02 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Menopause
Keywords: Menopause; Hot Flash; MENQOL; Mobile exercise device
MeSH Terms: conditions — Hot Flashes | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Active Comparator): This group will participate in a weekly exercise regimen and actively log the physical activity in a diary. They will complete the daily hot flash diary, MENQOL scale and calorimeter. All subjects will complete questionnaire (MENQOL Scale,) before the start of the study, at the sixth week of the study and after the completion of the twelfth week. A 2-week baseline assessment of hot flashes using the hot flash diary and fitbit flex will be followed by 12 weeks of assessment during the exercise intervention.
  Interventions: Behavioral: Exercise
- No Exercise (Active Comparator): They will complete the daily hot flash diary, MENQOL scale and calorimeter. All subjects will complete questionnaire (MENQOL Scale,) before the start of the study, at the sixth week of the study and after the completion of the twelfth week. A 2-week baseline assessment of hot flashes using the hot flash diary and fitbit flex will be followed by 12 weeks of assessment during the exercise intervention.
  Interventions: Behavioral: No exercise

INTERVENTIONS:
Behavioral: Exercise — Strength training exercises for older adults. All subjects will complete questionnaire (MENQOL Scale),hot flash diary and wear the fitbit flex for duration of study.
  Arms: Exercise Intervention
Behavioral: No exercise — All subjects will complete questionnaire (MENQOL Scale),hot flash diary and wear the fitbit flex for duration of study.
  Arms: No Exercise

SUMMARY:
A prospective randomized pragmatic trial will be used to obtain data on energy expenditure, temperature changes and vasomotor symptoms at baseline, during the intervention in which participants will be randomized to either exercise or to not exercise, and at the end of the 12-week intervention.

DETAILED DESCRIPTION:
During menopause, the main symptom that prompts women to seek medical attention is hot flashes. It is estimated that 75% of all menopausal women (approximately 50,000,000) will experience hot flashes, and that 15% will be severely affected. In addition to hot flashes, other significant climacteric symptoms include depression, insomnia, nervousness, fatigue, arthralgia, headache, vaginal dryness and night sweats. Most clinical trials assessing therapeutic efficacy use subjective reports (eg. questionnaires, diaries). The current gold standard for objective assessment of hot flashes is measuring the skin conductance level. However, there is still a relative discordancy between self reported and objectively detected hot flashes even with the use of skin conductance level. A combination of objective and subjective measures probably constitutes a valid assessment of vasomotor symptoms.

The menopausal transition is associated with a risk to increase in body weight and adiposity. Weight gain in the menopausal woman can be closely associated with aging but is also influenced by hormonal changes. Identifying modifiable factors that can prevent or attenuate theses changes is of great relevance. Resting energy expenditure decreases with age but also decreases with loss of ovarian function. There is little data on energy expenditure as it relates to the menopause and how influences such as exercise play a role in metabolic rate and how this may play a role in vasomotor symptoms. is an a portable monitor that will be used to collect minute by minute data on energy expenditure, physical activity and sleep monitoring. This data will be used to calculate temperature regulation. There are no studies using this device on women undergoing the menopause transition. Given the skin temperature fluxes that occur with hot flashes, it is possible that energy expenditure is not calculated correctly, since heat is used as a measure of energy expenditure. There are also no studies comparing this device to the current subjective evaluative methods like the hot flash diary and quality of life surveys. The purpose of this study is to generate preliminary data needed to conduct a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be women
* All subjects will be between the ages of 35 and 60
* Must experience 7-20, moderate-severe hot flashes/day or 50-140, moderate-severe hot flashes/week for greater than two months. Moderate or severe hot flashes are recurrent periods of heat sensation and sweating that either do not interfere with or cause the cessation of an activity, respectively
* Must have had a bilateral salpingo-oophorectomy for >12 months or amenorrhea >12 months
* Must have a signed informed consent
* Must be able to function independently in all activities of daily living and be capable of reliable documentation for at least six consecutive weeks.

Exclusion Criteria:

* Men and children will not be included.
* Have current history of fever, cough, dysuria or diarrhea (i.e., signs of infection).
* Have >10% of hot flashes predictably related to certain food ingestion alcohol intake.
* Have a history of "easily blushing" and have >10% hot flashes associated with embarrassing events or migraines.
* Have an MI, stroke, functional decline within 1 month.
* Have a history of somatoform disorder.
* Have an estimated creatinine clearance < 60ml/min.
* Fail to record data in the diary for >3 days during the 2 week baseline period.
* Unable or unwilling to make weekly visits over course of therapy
* Received any calcium channel antagonists or gabapentin for the past two weeks. Received estrogen, herbal estrogen, progestin, leuprolide acetate or tamoxifen within the past two months (if they would still like to participate, they will be required to undergo a 2 month washout period before enrolling in the study). Started clonidine, raloxifene or a new anti-depressant within the past month.
* Any contraindications to exercise or inability to exercise.
* Specific risks to resistance testing or training: Confirmed or suspected osteoporosis or osteopenia, musculo-skeletal injuries to involved joints, surgery within last year (includes eye surgery), hernia, Marfan syndrome, implanted pacemaker or defibrillator, low functional capacity (<4 METS), uncontrolled hypertension >160/100 mmHg represent a partial list of risks.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Change in hot flash rate occurrence with strength training exercise. | 12 weeks
  Hot Flash Diary, strength training manual and Fitbit flex will be used

SECONDARY OUTCOMES:
Hot Flash Diary | 14 weeks
  Measure Hot Flash duration and severity
Menopause-Specific Quality of Life Questionnaire (MENQOL) | 14 weeks
  Measure impact on daily life
Calorimeter | 14 weeks
  Measure basel metabolic rate
FitBit Data | 14 weeks
  Measure daily activity
Strength training log | 12 weeks
  Record strength training performed

CONTACTS AND LOCATIONS:
Overall Officials: Sireesha Y Reddy, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kronenberg F. Hot flashes: epidemiology and physiology. Ann N Y Acad Sci. 1990;592:52-86; discussion 123-33. doi: 10.1111/j.1749-6632.1990.tb30316.x. PMID 2197954
- [Background] Kass-Annese B. Alternative therapies for menopause. Clin Obstet Gynecol. 2000 Mar;43(1):162-83. doi: 10.1097/00003081-200003000-00018. PMID 10694998
- [Background] Guttuso TJ Jr. Gabapentin's effects on hot flashes and hypothermia. Neurology. 2000 Jun 13;54(11):2161-3. doi: 10.1212/wnl.54.11.2161. PMID 10851385
- [Background] Campbell S, Whitehead M. Oestrogen therapy and the menopausal syndrome. Clin Obstet Gynaecol. 1977 Apr;4(1):31-47. PMID 322905
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Reddy SY, Warner H, Guttuso T Jr, Messing S, DiGrazio W, Thornburg L, Guzick DS. Gabapentin, estrogen, and placebo for treating hot flushes: a randomized controlled trial. Obstet Gynecol. 2006 Jul;108(1):41-8. doi: 10.1097/01.AOG.0000222383.43913.ed. PMID 16816054
- [Background] Thurston RC, Sowers MR, Chang Y, Sternfeld B, Gold EB, Johnston JM, Matthews KA. Adiposity and reporting of vasomotor symptoms among midlife women: the study of women's health across the nation. Am J Epidemiol. 2008 Jan 1;167(1):78-85. doi: 10.1093/aje/kwm244. Epub 2007 Sep 19. PMID 17881385
- [Background] Tremollieres FA, Pouilles JM, Ribot CA. Relative influence of age and menopause on total and regional body composition changes in postmenopausal women. Am J Obstet Gynecol. 1996 Dec;175(6):1594-600. doi: 10.1016/s0002-9378(96)70111-4. PMID 8987946